CLINICAL TRIAL: NCT03876340
Title: Impact of a Clinical Decision Algorithm on Length of Hospital Stay and Costs of Care of Burned Patients: a Pragmatic Clinical Trial
Brief Title: Impact of a Clinical Decision Algorithm on Length of Hospital Stay and Costs of Care of Burned Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, MARIO AURELIO MARTÍNEZ-JIMÉNEZ, Chief of the Burn Unit, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QX2018
Record Dates: First submitted 2019-03-01; First posted 2019-03-15 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Burns
Keywords: Burns; Cost-effectiveness; Clinical decision rule; Length of stay; Cost of treatment
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Two parallel arms: group A will receive treatment as usual, group B will receive treatment as dictated by a clinical decision algorithm (PLoS ONE 2018:13(11):e0206477).
Who Masked: Participant, Outcomes Assessor
Masking Description: Controlled double blinded study. Patients and outcomes assessors will be masked to intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current treatment (Active Comparator): Patients will receive burn care treatment as dictated by the surgical team (current standard of care).
  Interventions: Other: Current treatment
- Algorithm-dictated treatment (Experimental): Patients will receive burn care treatment as dictated by the treatment algorithm (PLOS ONE 13(11): e0206477.).
  Interventions: Other: Treatment algorithm

INTERVENTIONS:
Other: Treatment algorithm — Digital infrared thermograms will be obtained during the first contact with the patients. Temperature recordings of the injured and healthy skin will be used to calculate the temperature difference between the structures. The thermograms will be used to dictate the initial treatment.
  Arms: Algorithm-dictated treatment
Other: Current treatment — Digital infrared thermograms will be obtained during the first contact with the patients. Temperature recordings of the injured and healthy skin will be used to calculate the temperature difference between the structures, but the results will be kept sealed until the study is finished. The patients will receive the usual standard of care as dictated by the surgical team.
  Arms: Current treatment

SUMMARY:
Reliable and valid assessment of burn wound depth or healing potential is essential to treatment decision-making, to provide a prognosis, and to compare studies evaluating different treatment modalities. Clinical evaluation remains the most widely used method for assessing the depth of the burn wound. This method is based on the subjective evaluation of visual and tactile characteristics of the wound, with an accuracy ranging between 50 to 70%; which is not precise to guide clinical decision making. The aim of these study is to validate thermography as a therapeutic approach to predict treatment modality based on thermographic imaging of the wound and its healing potential obtained during the first three days of treatment of either healing by re-epithelization, requiring skin grafts, or requiring amputations. By performing this algorithm, it is expected to address three aspects of the management of patients with acute burns: early clinical diagnosis, initial management decisions and reduction of hospitalization days.

DETAILED DESCRIPTION:
Burn wounds are divided into first degree burns involving the epidermis, superficial second degree with lesion of the papillary dermis, deep second degree with lesion of the reticular dermis, third degree with lesion to the hypodermis, and fourth degree involves fascia, muscle, tendons and bone.

In burns, development and severity of complications are in direct proportion to the magnitude of the burn. The magnitude of the damage depends on three factors, the duration of the contact, the intensity of the current or temperature and the resistance offered by the tissue. The extent of the burned skin surface is very useful to assess the severity of the patient, it is a relevant criterion to develop the prognosis. It is important to have comprehensive knowledge of the burned patient and close collaboration with the multidisciplinary care team through a careful evaluation that includes mechanism of injury, type, extent, degree of affectation and organic repercussion of the burn. The reliable and valid evaluation on the depth of a burn wound or the healing potential is essential for the decision making in the treatment; to provide a prognosis and to compare the different treatment modalities. There is no gold standard in the evaluation of burns.

Infrared imaging is a non-invasive technique that quantifies the temperature of the body surface by capturing the thermal radiation emitted and producing a high-resolution digital image called a thermogram. The presence of a disease interferes locally with the heat balance, which results in an increase or decrease in the temperature of the skin, in comparison to the surrounding regions or the contralateral not affected region. A degree of thermal asymmetry between opposite sides of the body (ΔT) of up to 1 ° C has been considered indicative of dysfunction. In several previous studies the parameters of initial thermography between the wound and healthy skin (delta T) were defined, to decide the therapeutic approach of the burns to predict the evolution: ΔT <3º C epithelialized with conservative treatment, ΔT 3-5º C should be graft early and ΔT> 5º C should be amputated.Thermography offers a feasible option for valuation.

Methods:

This is randomized clinical study of patients with different burn depth. All patients will be examined using a thermal camera.

Expected Results:

In all cases, the investigators obtained infrared images that corroborate clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partial or full thickness burn in <15% of the total body surface area in distal limbs, including hands or feet.
* Patients admitted to the burn care unit within 24 hours from injury.
* Patients that signed the informed consent. In the case of children or patients unable to consent themselves, signing of the consent by their guardian.

Exclusion Criteria:

* Patients who sustained electrical burns.
* Patients that received previous care in any other unit.
* Patients with uncontrolled chronic diseases.
* Patients that used corticosteroids or cytotoxic medications within 3 months of sustaining the injury.
* Patients with a baseline body mass index of <19.9 for adults or below the 5th percentile for their age in children.
* Presence of foreign bodies embedded in the wound tissue, gross edema, systemic causes of distal hypoperfusion, or presence of local infection.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | Through study completion, an average of 30 days
  Number of days the patient stays in the burn care unit
Treatment modality conversion | Through study completion, an average of 30 days
  Change of the initial treatment modality

SECONDARY OUTCOMES:
Rate of complications | Through study completion, an average of 30 days
  Presence of complications such as tissue necrosis, infection, death.
Cost of stay | Through study completion, an average of 30 days
  Total cost of the stay in the burn care unit in american dollars (USD)

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Ramirez Garcia Luna, MD, MSc, Study Chair — Universidad Autonoma de San Luis Potosi
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez-Jimenez MA, Ramirez-GarciaLuna JL, Kolosovas-Machuca ES, Drager J, Gonzalez FJ. Development and validation of an algorithm to predict the treatment modality of burn wounds using thermographic scans: Prospective cohort study. PLoS One. 2018 Nov 14;13(11):e0206477. doi: 10.1371/journal.pone.0206477. eCollection 2018. PMID 30427892
- [Background] Medina-Preciado JD, Kolosovas-Machuca ES, Velez-Gomez E, Miranda-Altamirano A, Gonzalez FJ. Noninvasive determination of burn depth in children by digital infrared thermal imaging. J Biomed Opt. 2013 Jun;18(6):061204. doi: 10.1117/1.JBO.18.6.061204. PMID 23111601
- [Background] Kolosovas-Machuca ES, Gonzalez FJ. Distribution of skin temperature in Mexican children. Skin Res Technol. 2011 Aug;17(3):326-31. doi: 10.1111/j.1600-0846.2011.00501.x. Epub 2011 Feb 22. PMID 21338404